CLINICAL TRIAL: NCT01137526
Title: A Randomized, Double-Blind, Placebo and Active-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ABT-384 in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety Study of ABT-384 in Subjects With Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M12-033; 2009 017801-12 (EudraCT Number)
Record Dates: First submitted 2010-05-07; First posted 2010-06-04 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(5-(aminocarbonyl)tricyclo(3.3.1.13,7)dec-2-yl)-alpha,alpha-dimethyl-4-(5-(trifluoromethyl)-2-pyridinyl)-1-piperazineacetamide; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ABT-384 Dose 1 (Experimental)
  Interventions: Drug: ABT-384
- ABT-384 Dose 2 (Experimental)
  Interventions: Drug: ABT-384
- donepezil (Active Comparator)
  Interventions: Drug: donepezil
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-384 — Subjects will take study drug once daily for 12 weeks
  Arms: ABT-384 Dose 1; ABT-384 Dose 2
Drug: donepezil — Subjects will take study drug once daily for 12 weeks.
  Other Names: Aricept
  Arms: donepezil
Drug: placebo — Subjects will take study drug once daily for 12 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to test if the investigational medication, ABT-384, is a safe and effective treatment for adults with mild-to-moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the safety and efficacy of ABT-384 in approximately 260 adults with mild-to-moderate Alzheimer's Disease (AD). Subjects will be randomized to one of four treatment groups (ABT-384, donepezil, or placebo) for a 12-week Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and caregiver must voluntarily sign and date and informed consent. If the subject is not fully competent, full informed consent must be obtained from a legal representative and assent must be obtained from the subject.
2. Subject is male or female between the ages of 55 and 90 years of age, inclusive, at Day-1.
3. Subject meets the NINCDS/ADRDA criteria for probable AD.
4. Subject has a Mini-Mental Status Examination (MMSE) score of 10 to 24, inclusive, at Screening Visit 1.
5. Subject has a Cornell Scale for Depression in Dementia (CSDD) score ≤ 10 at Screening Visit 1.
6. With the exception of a diagnosis of mild-to-moderate AD and the presence of stable medical conditions, the subject is generally in good health based on medical history, physical examination, vital signs, clinical lab tests and 12-lead ECG.
7. If female, subject must be postmenopausal for at least 2 years or surgically sterile.
8. If male, the subject is surgically sterile (vasectomy), is sexually inactive, or is using a barrier method of birth control.
9. Subject has an identified reliable, caregiver (e.g., family member, social worker, nurse), who will provide support and ensure compliance with the study medication and procedures.
10. Subject and caregiver are fluent in the language used for administration of the rating scales or cognitive tests and have sufficient visual, hearing and graphomotor skills to complete procedures.

Exclusion Criteria:

1. Subject has a known hypersensitivity or intolerance to donepezil that led to discontinuation or a known reported history of donepezil treatment failure.
2. Subject is currently taking or has taken a medication for the treatment of AD or dementia within 60 days of Screening Visit 1, or is participating in cognitive therapy for the treatment of AD or dementia.
3. Subject has a history of a drug or alcohol disorder (abuse/dependence), based on either DSM-IV-TR or ICD-10 criteria, excluding nicotine, within 2 years prior to Screening Visit 1.
4. In the opinion of the investigator, the subject has any clinically significant uncontrolled medical or psychiatric illness that would affect the safety of the subject.
5. The subject has a current thyroid disease or history of thyroid disease, and is not currently being treated with a stable dose of thyroid replacement medication.
6. For any reason the investigator considers the subject to be an unsuitable candidate to receive ABT-384 or donepezil.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to final observation in the Alzheimer's Disease Assessment Scale-Cognition portion (ADAS-cog) total score | 12 Weeks

SECONDARY OUTCOMES:
Mini Mental Status Examination (MMSE) score at Baseline, Weeks 4, 8, and 12 | 12 Weeks
Clinician's Interview Based Impression of Change-plus (CIBIC-plus) score at Baseline, Weeks 4, 8, and 12 | 12 Weeks
Neuropsychiatric Inventory (NPI) score at Baseline, Weeks 4, 8, and 12 | 12 Weeks
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score at Baseline, Weeks 4, 8, and 12 | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Marek, MD, Study Director — AbbVie
Locations (30):
- Russia (9):
  - Site Reference ID/Investigator# 36304, Kazan'
  - Site Reference ID/Investigator# 36306, Kirov
  - Site Reference ID/Investigator# 37944, Moscow
  - Site Reference ID/Investigator# 26904, Saint Petersburg
  - Site Reference ID/Investigator# 26902, Saint Petersburg
  - Site Reference ID/Investigator# 36305, Saint Petersburg
  - Site Reference ID/Investigator# 26909, Saratov
  - Site Reference ID/Investigator# 38383, Yaroslavl
  - Site Reference ID/Investigator# 40834, Yekaterinburg
- South Africa (3):
  - Site Reference ID/Investigator# 45584, Belville
  - Site Reference ID/Investigator# 47102, George
  - Site Reference ID/Investigator# 45583, Johannesburg
- Ukraine (9):
  - Site Reference ID/Investigator# 39855, Donetsk
  - Site Reference ID/Investigator# 26914, Kharkiv
  - Site Reference ID/Investigator# 26912, Kiev
  - Site Reference ID/Investigator# 40484, Lviv
  - Site Reference ID/Investigator# 27002, Poltava
  - Site Reference ID/Investigator# 39856, Poltava
  - Site Reference ID/Investigator# 40482, Simferopil
  - Site Reference ID/Investigator# 40483, Ternopil
  - Site Reference ID/Investigator# 35660, Vinnytsia
- United Kingdom (9):
  - Site Reference ID/Investigator# 36327, Bath
  - Site Reference ID/Investigator# 35657, Blackburn
  - Site Reference ID/Investigator# 36330, Crowborough
  - Site Reference ID/Investigator# 36326, Glasgow
  - Site Reference ID/Investigator# 44123, Ivybridge, Devon
  - Site Reference ID/Investigator# 35658, London
  - Site Reference ID/Investigator# 35902, Northampton
  - Site Reference ID/Investigator# 36328, Oxford
  - Site Reference ID/Investigator# 36329, Peterborough

REFERENCES:
- [Derived] Marek GJ, Katz DA, Meier A, Greco N 4th, Zhang W, Liu W, Lenz RA. Efficacy and safety evaluation of HSD-1 inhibitor ABT-384 in Alzheimer's disease. Alzheimers Dement. 2014 Oct;10(5 Suppl):S364-73. doi: 10.1016/j.jalz.2013.09.010. Epub 2014 Jan 10. PMID 24418055